CLINICAL TRIAL: NCT07131527
Title: Comparative Study Between the Efficacy of Pre- Operative Oral Gabapentin Versus Diclofenac Sodium in Post-operative Analgesia in Adult Undergoing Laparoscopic Cholecystectomy
Brief Title: Comparison Between Oral Gabapentin Versus Diclofenac Sodium in Post-operative Analgesia Laparoscopic Cholecystectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Manar Zakria Ismail, Resident , Anesthesia , Surgical Icu , Pain management Faculty of Medicine Sohag university, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Soh-Med--25-7-5MS
Record Dates: First submitted 2025-08-13; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Cholecystitis, Chronic
MeSH Terms: conditions — Cholecystitis; Bronchiolitis Obliterans Syndrome | interventions — Gabapentin; Diclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A will receive oral Gabapentin (Active Comparator): Patients included in this group will receive 600 mg of gabapentin 2 h before surgery.
  Interventions: Drug: Gabapentin
- group B will receive diclofenac sodium (Active Comparator): Patients included in this group will receive 100 mg diclofenac sodium 2 h before surgery.
  Interventions: Drug: Diclofenac Sodium

INTERVENTIONS:
Drug: Gabapentin — oral Gabapentin will be given 2 hours perioperative as postoperative analgesia patients undergoing laparoscopic cholecystectomy
  Arms: group A will receive oral Gabapentin
Drug: Diclofenac Sodium — oral diclofenac sodium will be given 2 hours perioperative as postoperative analgesia patients undergoing laparoscopic cholecystectomy
  Arms: group B will receive diclofenac sodium

SUMMARY:
this study amis to compare between perioperative oral Gabapentin versus Diclofenac sodium on postoperative analgesia patients undergoing laparoscopic cholecystectomy

ELIGIBILITY:
Inclusion Criteria:

Age from 20 to 60 years old. Both sexes. American Society of Anesthesiologists (ASA) physical status I- II. Patients undergoing laparoscopic cholecystectomy.

Exclusion Criteria:

Patients with hypertension. Pregnant women. Obese patients with BMI >35 kg/m2. Alcoholics. Patients With DM Patient refusal

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
the effect of preoperative oral Gabapentin versu Diclofenac sodium in adult patient undergoing laparoscopic cholecystectomy | 8 hours after operation
  postoperative pain by Numerical Rating Scale (0 represents "no pain" while 10 represents "the worst pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Egypt

REFERENCES:
- [Background] Abuahmed M, Rashid R. Day-case laparoscopic cholecystectomy in the management of gallbladder disease: a literature review. Langenbecks Arch Surg. 2024 Sep 28;409(1):292. doi: 10.1007/s00423-024-03479-6. PMID 39340655
- [Background] Nestor CC, Ng C, Sepulveda P, Irwin MG. Pharmacological and clinical implications of local anaesthetic mixtures: a narrative review. Anaesthesia. 2022 Mar;77(3):339-350. doi: 10.1111/anae.15641. Epub 2021 Dec 14. PMID 34904711
- [Background] LaForge JM, Urso K, Day JM, Bourgeois CW, Ross MM, Ahmadzadeh S, Shekoohi S, Cornett EM, Kaye AM, Kaye AD. Non-steroidal Anti-inflammatory Drugs: Clinical Implications, Renal Impairment Risks, and AKI. Adv Ther. 2023 May;40(5):2082-2096. doi: 10.1007/s12325-023-02481-6. Epub 2023 Mar 22. PMID 36947330